CLINICAL TRIAL: NCT03788330
Title: Effects of Fresh Air Filtration System on Indoor Air Quality and Children's Health in Shanghai Schools
Brief Title: Short-term Health Benefits of Using Fresh Air Filtration System in Classroom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhuohui Zhao, Investigation director, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: XFGY001
Record Dates: First submitted 2018-12-05; First posted 2018-12-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Airway Morbidity; Cognitive and Attention Disorders and Disturbances; Oxidative Stress
Keywords: exhaled nitric oxide; Sick building syndrome; indoor air
MeSH Terms: conditions — Cognition Disorders; Sick Building Syndrome | interventions — Filtration; Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fresh air system with filtration (Experimental): A fresh air ventilation system combined with PM2.5 filtration is applied in one primary school classroom.
  Interventions: Device: Fresh air system with filtration
- Fresh air system with no filtration (Placebo Comparator): A fresh air ventilation system with no PM2.5 filtration is applied in a parallel classroom.
  Interventions: Device: Fresh air system with filtration
- Natural ventilation (No Intervention): Natural ventilation system was applied in the 3rd classroom as normal.

INTERVENTIONS:
Device: Fresh air system with filtration — Using fresh air ventilation combined with PM2.5 filtration system to reduce the indoor PM2.5 concentration in primarty school classrooms
  Other Names: mechanical ventilation and filtration system
  Arms: Fresh air system with filtration; Fresh air system with no filtration

SUMMARY:
A randomized crossover trial will be conducted in 90 primary school children in 3 classrooms in Shanghai, China. The effects of fresh air ventilation/filtration system, fresh air ventilation system with no filtration and natual ventilation will be compared on the effects of reducing indoor PM2.5 and chilhood health. Biological samples of children are going to be collected to investigate the associations between indoor air pollution and biomarkes of certain health effects.

DETAILED DESCRIPTION:
A randomized crossover trial among 90 primary students in 3 classrooms in Shanghai, China will be performed. Three arms are going to be 1) fresh air filtration system, 2) fresh air system with no filtration and 3) natural ventilation. Each arm is going to be in use for five continuous weekdays followed by one week of wash-out. After one-week of wash out, a cross over change between 3 arms is going to be taked. Then the 2nd week of intervention is performed followed by the 2nd wash-out week. The same cross-over change between 3 arms is going to be repeated again until each classroom will be applied by all three arms of ventilation. A total of 5 weeks is required for the project. Children's biological samples including saliva, urine and skin samples will be collected as well as exhaled NO. A questionnaire on children's perception on air quality will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* All invited primary school children in Grade 5 in an artibrarily selected school

Exclusion Criteria:

* Current airway symptoms (cough, airway infection, asthma et al.)
* Acute infectious diseases

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide | within 2 hours of the end of intervention in each week
  Airway inflammation biomarker
Oxidative stress biomarkers | within 2 hours of the end of intervention in each week
  The level of lysozyme, cortisone and SIgA will be assessed in saliva and other oxidative biomarkers in the urine samples in children.
Sick building symdrom | within 2 hours of the end of intervention in each week
  Answering questionnaire on sick biulding symdrom

CONTACTS AND LOCATIONS:
Overall Officials: Zhuohui Zhao, Dr, Study Chair — Fudan University
Locations (1):
- Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No